CLINICAL TRIAL: NCT03975998
Title: Dutch-AMR Study: Early Mitral Valve Repair Versus Watchful Waiting in Asymptomatic Patients With Severe Organic Mitral Regurgitation and Preserved Ejection Fraction: a Multicenter Registry Trial
Brief Title: Dutch-AMR: Early Mitral Valve Repair Versus Watchful Waiting in Asymptomatic Patients With Severe Mitral Regurgitation
Acronym: Dutch-AMR
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Heart Institute (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amphia Hospital (Other); Maastricht University Medical Center (Other); Medisch Spectrum Twente (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, S.A.J. Chamuleau, MD, PhD, UMC Utrecht
Other Study IDs: 16/743
Record Dates: First submitted 2016-11-28; First posted 2019-06-05 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Mitral Regurgitation
Keywords: Mitral regurgitation; Mitral repair; Watchful waiting; Asymptomatic
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aymptomatic patients with severe mitral regurgitation: Watchful waiting Early Surgery
  Interventions: Procedure: Mitral valve repair

INTERVENTIONS:
Procedure: Mitral valve repair — Minimally invasive repair of severe organic mitral regurgiation

SUMMARY:
Rationale:

Severe asymptomatic organic Mitral Valve (MV) regurgitation with preserved left ventricular (LV) function is a challenging clinical entity as data on the recommended treatment strategy for these patients are scarce and conflicting, which is reflected in current guidelines. European guidelines advocate a more conservative strategy i.e. watchful waiting, with yearly echocardiography, whilst American guidelines are more in favour of early surgery to reconstruct the MV, i.e. MV repair (in contrast to MV replacement) in order to prevent future LV dysfunction and complaints.

A number of non-randomised trials show a favourable outcome of early surgery: in the study of Enriquez-Sarano et al. for instance, the early surgery strategy has shown to be associated with improved long-term survival, decreased cardiac mortality, and decreased morbidity compared with the conservative management [1]. On the other hand, non-randomised trials describe also that a conservative strategy (i.e. watchful waiting) can be safely accomplished. If facilitated surgery is performed in this population (50% at 10 years follow-up according to Rosenhek et al [2]), it has proven to be eventually associated with good perioperative and postoperative outcome when careful follow-up is being carried out [2].

Objective:

To compare early MV repair versus watchful waiting in asymptomatic patients with severe organic mitral valve regurgitation and preserved left ventricular function.

Study design:

Multicenter, registry trial.

Study population:

250 Asymptomatic patients (18-75 years old) with severe organic MV regurgitation and preserved left ventricular function. The current European Society of Cardiology (ESC) guidelines on Valvular Heart Disease will be applied [3]. These guidelines are also used in the Netherlands. Accordingly, patients with an indication for MV surgery will not be included.

Intervention:

Intervention will be early MV repair compared to a watchful waiting strategy.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years.
* Asymptomatic patients. "Asymptomatic" is defined as absence of subjective limitations of exercise capacity or complaints expressed by the patient and confirmed by the treating cardiologist.
* Severe organic mitral valve regurgitation. "Severe organic mitral valve regurgitation" is defined as non-ischemic mitral valve regurgitation with an organic cause (intrinsic valve lesion) as determined by echocardiographic core-lab reading based on the criteria for definition of severe MR as issued by the ESC guidelines [4]. For practical reasons, referring cardiologists can use an ESC guidelines based index that was validated in the investigator's core-lab (Jansen et al, Practical echocardiographic semi-quantitative scoring system to determine severity of mitral regurgitation. Abstract presentation at ESC EUROECHO Congress 2011 and annual spring congress 2012 Netherlands Society of Cardiology).
* Preserved left ventricular function, "Preserved left ventricular function" is defined as left ventricular ejection fraction >60% and left ventricular end-systolic dimension <45 mm (no indexed value, measured by echocardiography).
* The likelihood of MV repair should be more than 90% determined by the local heart team with a cardiologist and cardiothoracic surgeon.

Exclusion Criteria:

* Pulmonary hypertension (>50 mmHg at rest).
* Atrial fibrillation, either on 12-lead ECG or holter-monitoring.
* Physical inability as determined by the heart team to undergo surgery.
* Other life-threatening morbidity.
* Higher expected surgical risks in advance, according to the dedicated heart team.
* Patients with moderate to severe kidney disease (estimated glomerular filtration rate (eGFR) less than 30 mL/min).
* Flail leaflet together with a left ventricular end systolic diameter (LVESD) ≥40 mm (no indexed value)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic patients with severe organic mitral regurgitation and preserved ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Time to event: cardiovascular mortality, congestive heart failure, hospitalization, class I or class IIa indication for MV surgery | 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Amsterdam Medical Center (AMC), Amsterdam
  - Amphia Breda, Breda
  - Medisch Spectrum Twente (MST), Enschede
  - Leiden University Medical Center (LUMC), Leiden
  - Maastricht UMC, Maastricht
  - University Medical Center Utrecht (UMC Utrecht), Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ling LH, Enriquez-Sarano M, Seward JB, Orszulak TA, Schaff HV, Bailey KR, Tajik AJ, Frye RL. Early surgery in patients with mitral regurgitation due to flail leaflets: a long-term outcome study. Circulation. 1997 Sep 16;96(6):1819-25. doi: 10.1161/01.cir.96.6.1819. PMID 9323067
- [Background] Rosenhek R, Rader F, Klaar U, Gabriel H, Krejc M, Kalbeck D, Schemper M, Maurer G, Baumgartner H. Outcome of watchful waiting in asymptomatic severe mitral regurgitation. Circulation. 2006 May 9;113(18):2238-44. doi: 10.1161/CIRCULATIONAHA.105.599175. Epub 2006 May 1. PMID 16651470
- [Background] Vahanian A, Baumgartner H, Bax J, Butchart E, Dion R, Filippatos G, Flachskampf F, Hall R, Iung B, Kasprzak J, Nataf P, Tornos P, Torracca L, Wenink A; Task Force on the Management of Valvular Hearth Disease of the European Society of Cardiology; ESC Committee for Practice Guidelines. Guidelines on the management of valvular heart disease: The Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology. Eur Heart J. 2007 Jan;28(2):230-68. doi: 10.1093/eurheartj/ehl428. Epub 2007 Jan 26. No abstract available. PMID 17259184